CLINICAL TRIAL: NCT00200785
Title: Identification of the Antiplatelet Compounds of Garlic Ex Vivo
Brief Title: Identifying the Anti-Blood-Clotting Compounds in Garlic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Larry D. Lawson principal investigator, Silliker, Inc./Plant Bioactives Research Institute, Inc.
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: R21AT001512-01 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2010-01-11 (Estimated); Last update posted 2010-01-11 (Estimated); Status verified 2009-12

CONDITIONS: Arteriosclerosis; Intracranial Arteriosclerosis
Keywords: garlic
MeSH Terms: conditions — Arteriosclerosis; Intracranial Arteriosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Garlic powder in ambient water (Active Comparator): high allicin
  Interventions: Dietary Supplement: garlic powder added to ambient water
- garlic powder in boiling water (Experimental): no allicin
  Interventions: Dietary Supplement: garlic powder added to boiling water

INTERVENTIONS:
Dietary Supplement: garlic powder added to ambient water — consumed 2.7 grams of garlic powder added to ambient water (equivalent to 8 grams fresh or raw garlic) in a sandwich, once a day for four weeks
  Other Names: Global Marketing Assoc., Inc.
  Arms: Garlic powder in ambient water
Dietary Supplement: garlic powder added to boiling water — consumed 2.7 grams of garlic powder added to boiling water (equivalent to 8 grams of cooked garlic) in a sandwich, once a day for four weeks
  Other Names: Global Marketing Assoc., Inc.
  Arms: garlic powder in boiling water

SUMMARY:
This study will seek to identify the compound(s) in garlic that is (are) responsible for its ability to prevent the formation of blood clots (prevent platelet aggregation) and to determine the maximally effective dose and duration of the benefits. This study will also determine whether "cooked" garlic (garlic powder added to boiling water, no allicin present) is as effective as "fresh" garlic (garlic powder added to ambient water, high allicin present) and, if more than one compound is involved, and whether their combined effects are more significant than the effects of each compound alone.

DETAILED DESCRIPTION:
Published studies indicate that various types of undefined garlic products display antiplatelet activity. However, the compounds responsible for this antiplatelet effect have not been identified.

Acute studies. In acute (one day) studies, healthy participants will consume several doses of "fresh garlic" (garlic powder added to ambient water; up to the equivalent of 12 grams fresh garlic or 52 mg allicin) as a paste in a tuna sandwich. At 0, 2, 4, and 6 hours after consumption, the ability of platelets to aggregate in platelet-rich plasma (PRP) or in whole blood (WB), in response to a drug (collagen, ADP) that stimulates platelet aggregation, will be measured. After establishing the optimum dose and optimum time of the antiplatelet effect for each person, and if the effects are sufficiently strong, the effects of cooked garlic (garlic powder added to boiling water, no allicin present) and seven extracted fractions (oil, protein, fructans, etc.) will be determined, using the fractions at the same dose as their abundance in the established optimum dose of crushed fresh garlic.

Chronic studies. If only weak platelet effects are found for a high acute dose of "fresh" garlic, chronic studies will be conducted. In chronic studies, participants will consume 8.0 grams of "fresh garlic" (2.7 grams garlic powder added to ambient water, allicin content = 35 mg) as a paste in a tuna sandwich every day for four weeks and 8.0 grams of "boiled garlic" (2.7 grams garlic powder added to boiling water) in a sandwich every day for an additional four weeks, after a 1-week washout. The ability of platelets to aggregate in PRP and whole blood will be determined before and every week after garlic consumption begins and after the 1-week washout.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 19 to 30 kg/m2
* Plans to remain in the study area for the next year
* Willingness to abstain from nonsteroidal anti-inflammatory drugs (NSAID drugs for 1 week prior to each study test
* Willingness to abstain from consuming garlic and significant amounts of onion, chocolate, or purple grape juice for 3 days prior to each study test
* Willingness to participate in all study tests

Exclusion Criteria:

* Pregnancy or breast-feeding
* Serious medical condition
* Allergy to garlic or wheat
* Tobacco use
* Excessive alcohol consumption
* Under psychiatric care

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-03; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry D. Lawson, PhD, Principal Investigator — Silliker, Inc./Plant Bioactives Research Institute
Locations (1):
- Silliker, Inc./Plant Bioactives Research Institute, Orem, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: healthy participants were recruited in Utah county, Utah, in early 2006
Groups:
- Garlic Powder: High Allicin: garlic powder in ambient water
- Garlic Powder: No Allicin: garlic powder in boiling water
Period: First Intervention
Arm/Group | Garlic Powder: High Allicin | Garlic Powder: No Allicin
Started | 9 | 6
Completed | 9 | 6
Not Completed | 0 | 0
Period: Washout Period of 1 Week
Arm/Group | Garlic Powder: High Allicin | Garlic Powder: No Allicin
Started | 9 | 6
Completed | 9 | 6
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Garlic Powder: High Allicin | Garlic Powder: No Allicin
Started | 9 | 6
Completed | 9 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Garlic Powder: High Allicin | Garlic Powder: No Allicin | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 9 | 6 | 15.0
  >=65 years | 0 | 0 | 0.0
Age Continuous [Mean (Standard Deviation); unit: years] | 32.2 (13.7) | 36.5 (15.1) | 32.2 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7.0
  Male | 5 | 3 | 8.0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 6 | 15.0
electrical impedance (ohms) at 0 weeks [Mean (Standard Deviation); unit: ohms] — collagen-induced platelet aggregation in whole blood (WB)
  ohms | 12.7 (1.2) | 15.0 (1.6) | 13.9 (1.4)
percent platelet aggregation at 0 weeks [Mean (Standard Deviation); unit: percent platelet aggregation] — collagen-induced aggregation in platelet-rich plasma (PRP)
  percent platelet aggregation | 76.0 (1.6) | 71.8 (5.7) | 73.9 (3.7)

OUTCOME MEASURES:

1. Primary Outcome: Percent Platelet Aggregation
Description: percent platelet aggregation in collagen-induced platelet aggregation in platelet rich plasma (PRP)
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: percent platelet aggregation
Arm/Group | Garlic Powder: High Allicin | Garlic Powder: No Allicin
Number analyzed (Participants) | 9 | 6
percent platelet aggregation | 71.4 (4.3) | 72.5 (5.5)

2. Secondary Outcome: Electrical Impedance in Ohms
Description: Electrical impedance (ohms) was measured using 0.5 mL of whole blood plus 0.5 mL saline in a Chronolog Whole Blood aggregometer. Ten mL of whole blood were collected and tested every week. There is no mathematical correlation between impedance (ohms) and percent aggregation.
Time Frame: 4 weeks
Population: Nine persons participated in the "high allicin" test. Six of the same persons participated in the "no allicin" test.
Measure: Mean (Standard Deviation); unit: ohms
Arm/Group | Garlic Powder: High Allicin | Garlic Powder: No Allicin
Number analyzed (Participants) | 9 | 6
ohms | 13.8 (1.5) | 15.0 (1.5)

ADVERSE EVENTS:
Arm/Group | Garlic Powder: High Allicin | Garlic Powder: No Allicin
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6
Other Adverse Events (participants affected / at risk) | 0/9 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No